CLINICAL TRIAL: NCT06105853
Title: Towards Neurobehavioral Profiles and Models of Adaptive Stress Responses and Resilience in Individuals With Alcohol Use Disorder
Brief Title: Neurobehavioral Profiles of Adaptive Stress Responses in Individuals With Alcohol Use Disorder
Acronym: A03
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRR265-A03
Record Dates: First submitted 2023-09-14; First posted 2023-10-30 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder; Stress Reaction; Social Stress; Craving; Relapse; Addiction, Alcohol; Risk Behavior
Keywords: stress; resilience; craving; sensitization; habituation; cortisol; ecological momentary assessment; alcohol use disorder
MeSH Terms: conditions — Alcoholism; Fractures, Stress; Recurrence; Risk-Taking; Substance-Related Disorders | interventions — Psychological Tests

STUDY DESIGN:
Intervention Model Description: * longitudinal
  * multimodal
  * interventional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): All participants will be exposed to the Trier Social Stress Test, followed by an alcohol cue-exposure in a barlab environment and functional magnetic resonance imaging assessing neural alcohol cue-reactivity, inhibition performance, emotion processing and resting state functional connectivity twice on two consecutive days.
  Interventions:
  Behavioral: Trier Social Stress Test
  Behavioral: Cue-Exposure to the favorite drink in a barlab setting
  Interventions: Behavioral: Trier Social Stress Test; Behavioral: Barlab Cue-Exposure; Behavioral: Functional magnetic resonance imaging

INTERVENTIONS:
Behavioral: Trier Social Stress Test — Test to induce high levels of acute social stress, including actors, representing the judging panel, and a faked exam situation (15 minutes duration).
Behavioral: Barlab Cue-Exposure — Participants are exposed to a bar situation with their individual favorite alcohol presented. They handle their favorite alcoholic drink and water (9 minutes duration).
Behavioral: Functional magnetic resonance imaging — Participants undergo a fMRI screening including three different behavioral tasks assessing alcohol cue reactivity, response inhibition, and emotion processing

SUMMARY:
The goal of this observational study is to investigate longitudinal stress response profiles and adaptive versus non-adaptive stress responses in alcohol use disorder. The main questions the projects aims to answer are:

What are the neurobehavioral underpinnings of adaptive stress responses and resilience to repeated stress exposure with regards to:

* alcohol craving?
* alcohol use?
* their modulation by prior stress exposure, social interactions, coping strategies and individual health behavior?

Participants will:

* be exposed to an established experimental stress-induction protocol, the Trier Social Stress Test
* be exposed to their favorite drink in a bar lab environment
* be assessed using fMRI to determine their neural alcohol cue reactivity, response inhibition, and emotion processing
* conduct an ambulatory phase to assess stressors, alcohol craving, substance use and details on social interactions, health behavior and coping strategies using ecological momentary assessment tools.

DETAILED DESCRIPTION:
The main objective of the study is to identify longitudinal profiles and models of adaptive stress responses and stress resilience in individuals with alcohol use disorder (AUD) and understand how stress and different responses to it influence alcohol craving and alcohol use trajectories over time. To achieve these goals, the investigators will examine habituation vs. sensitization of cortisol responses to repeated experimental stress exposure in individuals with AUD, as an established experimental model to studying adaptive vs. non-adaptive stress responses in the framework of an experimental set-up including an initial rest period (30 minutes), followed by the Trier Social Stress Test (15 minutes), exposure to the favorite drink in a bar environment (9 minutes) and functional magnetic resonance imaging (75 minutes) assessing A) neural alcohol cue-reactivity, B) inhibition performance during a Stop Signal Task, C) emotion processing during a face-matching task and D) resting state connectivity. The investigators also seek to characterize the neurobehavioral underpinnings of sensitized vs. habituated responses to repeated stress exposure, using an established alcohol cue-reactivity fMRI paradigm, and determine the impact of sensitized vs. habituated stress responses on physiological and subjective stress markers, alcohol craving, alcohol use, as well as their modulation by prior stress exposure, social support, drinking goals and individual health behavior with a focus on potentially modifiable factors that could serve as targets for future ecological momentary interventions. This setup will be repeated on a second examination day.

In addition, the investigators aim to assess whether the observed habituation vs. sensitization phenotypes to repeated stress exposure translate into everyday-life of the respective individual and predict adaptive vs. non-adaptive stress responses. To this end, the investigators will acquire ambulatory assessments with high temporal resolution over six weeks, including detailed mapping of exposure to micro- and macro-stressors, drinking motifs, alcohol craving, alcohol use and data on factors that potentially modify the association between stress and alcohol use, such as social interactions, stress coping strategies, drinking goals and individual health behavior (e.g., sleep, physical activity) to assess whether the observed habituation vs. sensitization phenotypes to repeated stress exposure translate into everyday-life of the respective individual and predict real-life stress responses and alcohol use.

Study flow:

Screening (telephone): Assessing study eligibility

Experimental study visit 1: Rest period (30 minutes) - Trier Social Stress Test (15 minutes) - Alcohol cue exposure (9 minutes) - fMRI (75 minutes)

Experimental study visit 2: Repetition of setup from 'experimental study visit 1'

Following six weeks: Ambulatory phase (smartphone tool) with daily requests regarding stressors, alcohol craving and consumption as well as health behavior

ELIGIBILITY:
Inclusion criteria are:

* age between 16 and 65 years
* meeting at least 2 criteria of an alcohol use disorder according to the Diagnostic and Statistical Manual of Mental Disorders (Fifth Edition) (DSM-5), yet without the need for a therapeutic intervention
* fluency in German
* able to understand the study procedures and give informed consent
* willingness to use a study smartphone

Exclusion criteria are:

* current use of drugs or medications that interact with the central nervous system or the glucocorticoid system
* contraindications for magnetic resonance imaging
* medical history of bipolar disorder, psychotic disorder, schizophrenia or schizophrenic spectrum disorder, or substance use disorder other than alcohol, nicotine, or cannabis
* medical history of severe head injury or other severe central nervous system disorders or other severe somatic disorders (e.g. liver cirrhosis)
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Cortisol | Assessed at 4 time points at each examination day: after a 30-minute rest period [0:30 hours]; after the 15-minute stress intervention [0:45 hours]; after the 9-minute Barlab exposure [0:54 hours]; after the 75-minute fMRI [2:09 hours]
  Cortisol levels measured in saliva as a stress marker (in nmol/l)
Alcohol urges | Assessed at 4 time points at each examination day: after a 30-minute rest period [0:30 hours]; after the 15-minute stress intervention [0:45 hours], after the 9-minute Barlab exposure [0:54 hours]; after the 75-minute fMRI [2:09 hours]
  self-report questionnaire: "Alcohol Urge Questionnaire (AUQ)" with Bohn et al. 1995; containing 8 items; each item will be rated on a 7-point-Likert-Scale from 1 "not true at all" (minimum) to 7 "completely true" (maximum); sum score is defined as outcome and higher outcome reflects higher alcohol urges
Alcohol craving | Assessed at 4 time points at each examination day: after a 30-minute rest period [0:30 hours]; after the 15-minute stress intervention [0:45 hours]; after the 9-minute Barlab exposure [0:54 hours]; after the 75-minute fMRI [2:09 hours]
  self-report "How strong is your craving for alcohol?"; containing 1 item; reported on a visual analogue scale ranging from 0 ("no craving") to 100 ("very strong craving")
Subjective stress level | Assessed at 4 time points at each examination day: after a 30-minute rest period [0:30 hours]; after the 15-minute stress intervention [0:45 hours]; after the 9-minute Barlab exposure [0:54 hours]; after the 75-minute fMRI [2:09 hours]
  self-report questionnaire: "Primary Appraisal Secondary Appraisal (PASA)"; Gaab, 2009; containing 16 items; each item will be rated on a 6-Point-Scale from 1 ("completely wrong") to 6 ("quite right"); sum score is defined as outcome and higher outcome reflects a higher subjective stress level
Neural alcohol-related cue-reactivity | at examination day: after 1:00 hour of the experimental procedure
  percent signal change from baseline condition (i.e. fixation cross), measured with fMRI; paradigm Vollstädt-Klein et al. 2010; [percent signal change is not a change over time; it is measured during one experimental session]; presentation of neutral and alcoholic (categories: beer, wine, spirits) stimuli in 20 blocks (blocked design; one block à 5 stimuli each presented for 4 seconds), after each block participants had to rate their craving: "I have alcohol craving." from 0 ("no craving at all") to 100 ("severe craving"), maximum rating duration is 10 seconds, following the rating a fixation cross was presented (10 seconds), total task duration: 12 minutes
Neural inhibition processing | at examination day: after 1:00 hour of the experimental procedure
  percent signal change from baseline condition (i.e. fixation cross), measured with fMRI; stop-signal reaction time task (Fauth-Buhler et al. 2012) [percent signal change is not a change over time; it is measured during one experimental session]; conduction of a stop-signal task of 600 trials (500 go-trials and 100 stop trials, participant have to respond as quickly as possible by pressing the left or right button according to the arrow direction, between the trials a fixation cross was presented (for 700 milliseconds to 1100 milliseconds), total task duration: 19 minutes
Neural emotion processing | at examination day: after 1:00 hour of the experimental procedure
  percent signal change from baseline condition (i.e. fixation cross), measured with fMRI; faces task (Hariri et al. 2002) [percent signal change is not a change over time; it is measured during one experimental session]; participants were exposed to faces with varying emotions and forms (geometric shapes as a sensorimotor control task) and had to match one of two simultaneously presented images with an identical target image, a total of nine blocks (four with faces, five controls) each lasting 32 seconds and a total duration of about five minutes
Resting state activity | at examination day: after 1:00 hour of the experimental procedure
  resting state connectivity measured with fMRI
Ecological momentary assessment | starting at the examination day until 6 weeks later; daily requests
  Self-report ratings of: Real-life alcohol craving with the item "How strong is your current alcohol craving?", rating with a 7-Point-Likert-Scale from 1 "no craving" to 7 "extreme craving"; of stress exposure with the item "How strong is your current level of stress?", rating with a 7-Point-Likert-Scale from 1 "not at all" to 7 "very stressed"; of alcohol consumption with the item "Remember yesterday: Which and how many alcoholic drinks did you consume?", a short-list with listed drinks and amounts will open from which participants can choose; and of stress coping with the item "How did you deal with unpleasant situations since the last prompt?", rating with a 5-Point-Likert-Scale from 1 "not at all" to 5 "excellent"

SECONDARY OUTCOMES:
Blood pressure (systolic and diastolic) | Assessed at 4 time points at each examination day: after a 30-minute rest period [0:30 hours]; after the 15-minute stress intervention [0:45 hours]; after the 9-minute Barlab exposure [0:54 hours]; after the 75-minute fMRI [2:09 hours]
  acquired with pressure sleeve (in mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Bach, MD, PhD, Principal Investigator — Central Institute of Mental Health; Falk Kiefer, MD, Principal Investigator — Central Institute of Mental Health; Clemens Kirschbaum, PhD, Principal Investigator — Technical University Dresden
Locations (2):
- Germany (2):
  - Central Institute of Mental Health, Mannheim, Baden-Wurttemberg
  - Central Institute of Mental Health, Mannheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fauth-Buhler M, de Rover M, Rubia K, Garavan H, Abbott S, Clark L, Vollstadt-Klein S, Mann K, Schumann G, Robbins TW. Brain networks subserving fixed versus performance-adjusted delay stop trials in a stop signal task. Behav Brain Res. 2012 Nov 1;235(1):89-97. doi: 10.1016/j.bbr.2012.07.023. Epub 2012 Jul 20. PMID 22820235
- [Background] Kirschbaum C, Prussner JC, Stone AA, Federenko I, Gaab J, Lintz D, Schommer N, Hellhammer DH. Persistent high cortisol responses to repeated psychological stress in a subpopulation of healthy men. Psychosom Med. 1995 Sep-Oct;57(5):468-74. doi: 10.1097/00006842-199509000-00009. PMID 8552738
- [Background] Bohn MJ, Krahn DD, Staehler BA. Development and initial validation of a measure of drinking urges in abstinent alcoholics. Alcohol Clin Exp Res. 1995 Jun;19(3):600-6. doi: 10.1111/j.1530-0277.1995.tb01554.x. PMID 7573780
- [Background] Gaab J. PASA - Primary Appraisal Secondary Appraisal. Verhaltenstherapie. 2009; 114-115.
- [Background] Hariri AR, Tessitore A, Mattay VS, Fera F, Weinberger DR. The amygdala response to emotional stimuli: a comparison of faces and scenes. Neuroimage. 2002 Sep;17(1):317-23. doi: 10.1006/nimg.2002.1179. PMID 12482086
- [Background] Vollstadt-Klein S, Wichert S, Rabinstein J, Buhler M, Klein O, Ende G, Hermann D, Mann K. Initial, habitual and compulsive alcohol use is characterized by a shift of cue processing from ventral to dorsal striatum. Addiction. 2010 Oct;105(10):1741-9. doi: 10.1111/j.1360-0443.2010.03022.x. PMID 20670348
- [Background] Bach P, Reinhard I, Koopmann A, Bumb JM, Sommer WH, Vollstadt-Klein S, Kiefer F. Test-retest reliability of neural alcohol cue-reactivity: Is there light at the end of the magnetic resonance imaging tube? Addict Biol. 2022 Jan;27(1):e13069. doi: 10.1111/adb.13069. Epub 2021 Jun 15. PMID 34132011